CLINICAL TRIAL: NCT01555164
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Ranolazine When Added to Metformin in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Phase 3 Study of Ranolazine in Subjects With Type 2 Diabetes Who Are Inadequately Controlled on Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-259-0147; 2012-001259-37 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine; Metformin; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine+metformin (Experimental): Qualifying Period: Participants will receive metformin 1000 mg + placebo to match ranolazine twice daily for either 2 or 8 weeks (dependent on metformin dose and HbA1c level at Screening).
  Treatment Period: Participants will receive ranolazine 500 mg + metformin 500 mg + placebo to match metformin twice daily on Days 1 through 7, followed by ranolazine 1000 mg + metformin 500 mg + placebo to match metformin twice daily from Day 8 through Week 24.
  Participants are required to maintain their diet and exercise regimen.
  Interventions: Drug: Ranolazine; Drug: Metformin; Drug: Placebo to match metformin; Behavioral: Diet; Behavioral: Exercise
- Placebo+metformin (Placebo Comparator): Qualifying Period: Participants will receive metformin 1000 mg + placebo to match ranolazine twice daily for either 2 or 8 weeks (dependent on metformin dose and HbA1c level at Screening).
  Treatment Period: Participants will receive metformin 1000 mg + placebo to match ranolazine twice daily through Week 24.
  Participants are required to maintain their diet and exercise regimen.
  Interventions: Drug: Placebo to match ranolazine; Drug: Metformin; Behavioral: Diet; Behavioral: Exercise

INTERVENTIONS:
Drug: Ranolazine — Ranolazine tablet(s) administered orally
  Other Names: Ranexa®
  Arms: Ranolazine+metformin
Drug: Placebo to match ranolazine — Placebo to match ranolazine for the duration of the study
  Arms: Placebo+metformin
Drug: Metformin — Metformin tablet(s) administered orally once daily
Drug: Placebo to match metformin — Placebo to match metformin for the duration of the study
  Arms: Ranolazine+metformin
Behavioral: Diet — Participants are instructed to continue the diet regimen prescribed by their physician.
Behavioral: Exercise — Participants are instructed to continue the exercise regimen prescribed by their physician.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to determine the effect of ranolazine when added to metformin on glycemic control in adults with type 2 diabetes mellitus (T2DM) who are inadequately controlled despite current treatment with stable metformin therapy in addition to diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of T2DM
* Metformin therapy at a stable total daily dose ≥ 1500 mg and ≤ 2550 mg in addition to diet and exercise for ≥ 8 weeks prior to Screening
* Body mass index (BMI) 25 to 45 kg/m^2, inclusive, at Screening
* HbA1c within specified ranges at Screening and at the end of the Qualifying Period based on current metformin dose
* C-peptide ≥ 0.8 ng/mL at Screening
* Fasting serum glucose (FSG) ≥ 130 mg/dL (7.2 mmol/L) and ≤ 240 mg/dL (13.3 mmol/L) at Screening and at the end of the Qualifying Period

Exclusion Criteria:

* Type 1 diabetes mellitus
* History of diabetic ketoacidosis, ketosis-prone diabetes, or hyperosmolar hyperglycemic coma
* History of severe hypoglycemia
* Any clinically significant cardiovascular or cerebrovascular event ≤ 3 months prior to Screening
* History of congestive heart failure
* Corrected QT interval (QTc) > 500 msec by ECG at Screening, a personal or family history of QTc prolongation, congenital long QT syndrome, or individuals who are receiving drugs that prolong the QTc interval, such as Class Ia or Class III antiarrhythmic agents, erythromycin, and certain antipsychotics (eg, ziprasidone)
* Serum creatinine concentration ≥ 1.5 mg/dL for males or ≥ 1.4 mg/dL for females at Screening
* Active liver disease and/or significant abnormal liver function defined as aspartate aminotransferase (AST) > 3 x upper limit of the normal range (ULN) and/or alanine aminotransferase (ALT) > 3 x ULN and/or serum total bilirubin > 2.0 mg/dL
* Use of any non-insulin antihyperglycemic therapy (other than metformin) for more than 14 days (consecutive or not) during the 12 weeks (24 weeks for thiazolidinediones) prior to Screening and/or use of any antihyperglycemic therapy other than metformin, at any dose, at any time during the 4 weeks prior to randomization
* Treatment with chronic insulin within 24 weeks prior to Screening (except for one temporary period of daily insulin injections no longer than 7 days)
* Treatment with strong or moderate cytochrome P450 3A (CYP3A) inhibitors or P-glycoprotein (P-gp) inhibitors within 14 days prior to randomization
* Treatment with CYP3A inducers or P-gp inducers within 14 days prior to randomization
* Treatment with simvastatin or lovastatin at a dose > 20 mg or > 40 mg daily, respectively, within 14 days prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yue, MD, Study Director — Gilead Sciences
Locations (146):
- United States (60):
  - Fundamental Research LLC, Gulf Shores, Alabama
  - KLR Business Group DBA Arkansas Clinical Research, Little Rock, Alaska
  - Radiant Research, Inc., Chandler, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Clinical Research Advantage, Tempe, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - National Research Institute, Los Angeles, California
  - Ritchken and First MD's, San Diego, California
  - Clearview Medical Research, LLC, Santa Clarita, California
  - Metabolic Institute of America, Tarzana, California
  - University Clinical Investigators, Tustin, California
  - Infosphere Clinical Research, West Hills, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Boca Raton Clinical Research Associates, Inc., Boca Raton, Florida
  - MD Clinical Institute, Hallandale, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Florida Institute for Clinical Research LLC, Orlando, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - Synergy Therapeutic Partners, Atlanta, Georgia
  - Perimeter Institute for Clinical Research, Atlanta, Georgia
  - Columbus Research Foundation, Columbus, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Choose To Lose, Eagle, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Covington Medical Care, Mandeville, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - Bellevue Family Practice, Bellevue, Nebraska
  - Clinical Research Advantage, Henderson, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - PhysiqueMed Clinical Trials, Greensboro, North Carolina
  - Clinical Trials of America Inc, Hickory, North Carolina
  - University Medical Associates, Huntersville, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Carolina Research Center, Shelby, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Rapid Medical Research, Inc, Cleveland, Ohio
  - Columbus Clinical Research Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Blair Medical Associates Inc., Altoona, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Holston Medical Group, P.C., Bristol, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Corpus Christi, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - West Houston Clinical Research, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Juno Research, LLC, Katy, Texas
  - Northeast Clinical Research of San Antonio, LLC, Schertz, Texas
  - Sugarland, Texas
  - Progressive Clinical Research, LLC, Bountiful, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Burke Internal Medicine, Inc., Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
- Canada (4):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Diabetes Research Clinic, Vancouver, British Columbia
  - Joanne F. Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - Source Unique Research, Hawkesbury, Ontario
- Czechia (2):
  - Nemocnice s poliklinikou Havirov, Havířov, Moravskoslezský kraj
  - Restrial s.r.o., Prague, Prague
- Hungary (5):
  - Synexus Hungary Ltd, Budapest
  - Selye János Kórház és Rendel?intézet, Belgyógyászati Szakrendelés, Komárom
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Medifarma 98, Nyíregyháza
  - Borbanya Praxis Kft., Outpatient Clinic, Nyíregyháza
- India (22):
  - Diabetomics India, Hyderabad, Andhra Pradesh
  - DHL Research Centre, 2nd Floor, Ahmedabad, Gujarat
  - Dia Care- A Complete Diabetes Care Center, Ahmedabad, Gujarat
  - Baroda Medical College and SSG Hospital, Vadodara, Gujarat
  - Banker's Heart Institute, Vadodara, Gujarat
  - Endocrinology & Diabetes Research Centre, Bangalore, Karnataka
  - Manipal Hospital, Bangalore, Karnataka
  - Endocrinology Diabetes Centre, Bangalore, Karnataka
  - Bangalore Diabetes Hospital, Bangalore, Karnataka
  - The Bangalore Diabetes Hospital, Bangalore, Karnataka
  - Jnana Sanjeevani Medical Center, Bangalore, Karnataka
  - Vinaya Hospital and Research Centre, Mangalore, Karnataka
  - Seth G. S. Medical College and KEM Hospital, Mumbai, Maharashtra
  - Institue of Clinical Endocrinology (I.C.E) and Diabetes Care Unit (D.C.U),, Nagpur, Maharashtra
  - Getwell Hospital and Research Institute, Nagpur, Maharashtra
  - Diabetes Care and Research Centre, Pune, Maharashtra
  - KEM Hospital Research Center, Pune, Maharashtra
  - Fortis City Centre, Chandigarh, Punjab
  - Diabetes and Heart Centre, Ludhiana, Punjab
  - Swamy Diabetes Centre, Chennai, Tamil Nadu
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Centre & Hospital, Coimbatore, Tamil Nadu
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Edith Wolfson Medical Center, Holon
  - Ziv Medical Center Safed-Israel, Safed
- Instituto Jalisciense de Investigación en Diabetes y Obesidad, Guadalajara, Jalisco, Mexico
- Poland (4):
  - LANDA - Specjalistyczne Gabinety Lekarskie, Krakow, Lesser Poland Voivodeship
  - Niepubliczy Zaklad Opieki Zdrowotnej (NZOZ) Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok
  - NZOZ "Esculap" S.C., Gniewkowo
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Sp. Komandytowo - Akcyjna, Lodz, Łódź Voivodeship
- Russia (25):
  - GOU VPO "Chita State Medical Academy" of Minzdravsocrazvitie RF, Chita
  - Clinic of New Medical Technology Company Limited, Dzerzhinskiy
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - State Institution of Public Health of Moscow City Endocrinology Dispensary, Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - Reafan, LLC, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University, Ryazan
  - Medinet, LLC, Saint Petersburg
  - North-Western State Medical Unversity n.a. I.I.Mechnikov, Saint Petersburg
  - Saint-Petersburg City Outpatient Clinic#37, Saint Petersburg
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - City Diabetology Center #4, "City Polyclinic #77", Saint Petersburg
  - Alexanders City Hospital, Saint Petersburg
  - Clinical Hospital #122 n.a. Sokolov of FMBA, Saint Petersburg
  - ANO Medical Centre XXI Century, Saint Petersburg
  - City Hospital #38 named after N. A. Semashko, Saint Petersburg
  - Krestovsky Island Medical Institute, LLC, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology named after V.A. Almazov, Saint Petersburg
  - Federal State Budget Military Educational Institution Medical Military Academy n. a. S. M. Kirov, Saint Petersburg
  - SPb GBUZ Diagnostic Center #85, Saint Petersburg
  - Center "Diabetes", LLC, Samara
  - Smolensk State Medical Academy, Sanatorium-Preventorium, Smolensk
  - City Hospital named after N.A.Semashko, Yaroslavl
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- South Africa (10):
  - Vawda Z Private Practice, Kwa Zulu Natal, Durban
  - Centre for Diabetes and Endocrinology Suite 1, KwaKhangela, Durban
  - Newkwa Medical Centre, Newlands West, Durban
  - Drs. Naiker and Naicker Inc., Overport, Durban
  - Synexus Clinical Research SA (Pty) Ltd, Meyerspark, Pretoria
  - East Rand Research Trading as Worthwhile Clinical Trials, Benoni
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Aliwal Shoal Medical & Clinical Trial Centre, Kwa Zulu Natal
  - Netcare Umhlanga Medical Centre, Kwa Zulu Natal
  - Helderberg Clinical Trials Centre, Somerset West
- Ukraine (10):
  - Educational Scientific Medical Centre, Donetsk National Medical University, Donetsk
  - State Institution "Institute of Problems of Endocrine Pathology n.a. V.Y. Danylevsky of NAMS of Ukra, Kharkiv
  - Ukrainian Scientific-and-Practical Center of Endocrine Surgery, Transplantation of Endocrine Organs, Kyiv
  - Department of Endocrinology of Railway Clinical Hospital #2 of station "Kyiv" of South East Railroad, Kyiv
  - Administration of Medical Service and Rehabilitation of "ARTEM" State Holding Company, Kyiv
  - National Medical University n.a. O.O. Bogomolets, Chair of Family Medicine based on Outpatient Clini, Kyiv
  - V. P. Komissarenko Institute of Endocrinology and Metabolism of AMS of Ukraine, Kyiv
  - Odessa State Medical University, Odesa
  - Odessa City Policlinic #20, Odesa
  - Vinnytsya Regional Clinical Endocrinology Dispensary, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled (during the Qualifying Period) at a total of 112 study sites in Canada, Europe, Asia, Mexico, South Africa, and the United States. The first participant was screened on 28 June 2012. The last participant observation occurred on 01 October 2013.
Pre-assignment Details: 580 participants entered the qualifying period; 442 participants were randomized and treated, and comprise the Safety Analysis Set. Of these, 20 participants were excluded due to major eligibility criteria protocol violation or because the participant had no postbaseline data; the remaining 422 participants comprise the Full Analysis Set.
Groups:
- Placebo+Metformin: Qualifying period: Metformin 1000 mg (2 x 500 mg tablets) twice daily plus placebo to match ranolazine twice daily for either 2 or 8 weeks (dependent on metformin dose and HbA1c level at Screening) and participants who were ≥ 80% compliant and meeting eligibility criteria continued to the treatment period.
  Treatment period: Metformin 1000 mg (2 x 500 mg tablets) twice daily plus placebo to match ranolazine twice daily through Week 24.
  Participants were required to maintain their diet and exercise regimen.
- Ranolazine+Metformin: Qualifying period: Metformin 1000 mg (2 x 500 mg tablets) twice daily plus placebo to match ranolazine twice daily for either 2 or 8 weeks (dependent on metformin dose and HbA1c level at Screening) and participants who were ≥ 80% compliant and meeting eligibility criteria continued to the treatment period.
  Treatment period: Ranolazine 500 mg (1 x 500 mg tablet) twice daily plus metformin 500 mg/metformin placebo (1 x 500 mg tablet active metformin plus 1 placebo tablet) twice daily on Days 1 through 7, followed by ranolazine 1000 mg (2 x 500 mg tablets) twice daily plus metformin 500 mg/metformin placebo (1 x 500 mg tablet active metformin plus 1 placebo tablet) twice daily from Day 8 through Week 24.
  Participants were required to maintain their diet and exercise regimen.
Period: Overall Study
Arm/Group | Placebo+Metformin | Ranolazine+Metformin
Started | 222 | 220
Completed | 182 | 185
Not Completed | 40 | 35
Not completed — Adverse Event | 5 | 7
Not completed — Hyperglycemia | 0 | 1
Not completed — Investigator's Discretion | 2 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 9 | 5
Not completed — Subject Non-compliance | 14 | 6
Not completed — Subject Withdrew Consent | 6 | 11

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Metformin | Ranolazine+Metformin | Total
Number analyzed (Participants) | 222 | 220 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8.9) | 56 (9.3) | 56 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 121 | 219
  Male | 124 | 99 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 37 | 90
  Not Hispanic or Latino | 166 | 181 | 347
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 52 | 54 | 106
  Black or African American | 8 | 11 | 19
  White | 160 | 153 | 313
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 82 | 67 | 149
  Hungary | 8 | 8 | 16
  Czech Republic | 0 | 1 | 1
  Mexico | 6 | 4 | 10
  Canada | 1 | 3 | 4
  Poland | 0 | 5 | 5
  Ukraine | 35 | 29 | 64
  South Africa | 7 | 4 | 11
  Israel | 2 | 1 | 3
  Russian Federation | 37 | 49 | 86
  India | 44 | 49 | 93
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (4.46) | 31.6 (4.95) | 31.4 (4.71)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 90.8 (20.01) | 89.9 (21.82) | 90.4 (20.91)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c in blood] | 8.09 (0.729) | 8.10 (0.692) | 8.09 (0.710)
Fasting Serum Glucose (FSG) [Mean (Standard Deviation); unit: mg/dL] | 170.0 (35.97) | 168.8 (32.86) | 169.4 (34.42)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.7 (5.31) | 6.4 (5.37) | 6.5 (5.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: The average (mean) change from baseline in HbA1c at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set (randomized participants who received ≥ 1 dose of study treatment with a baseline and at least one postbaseline measurement of HbA1c, excluding participants with major eligibility violations, and analyzed based on randomized treatment, regardless of actual treatment received) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent of HbA1c in blood
Arm/Group | Placebo+Metformin | Ranolazine+Metformin
Number analyzed (Participants) | 174 | 179
percent of HbA1c in blood
  HbA1c at Week 24 | 7.86 (1.003) | 7.72 (1.069)
  Change from baseline in HbA1c at Week 24 | -0.20 (0.949) | -0.37 (0.916)
Statistical Analysis 1: Comparison: Placebo+Metformin vs Ranolazine+Metformin; Assuming a common standard deviation of 1.2%, an effective sample size of 400 would provide at least 90% power to detect a statistically significant treatment difference of -0.4% (ranolazine vs. placebo) for the reduction of HbA1c from baseline at Week 24 based on a 2-sided alpha of 0.05 and 1:1 randomization; Test type: Superiority or Other; p = 0.306, Mixed Effects Model Analysis — P-value from a mixed-effect model including terms for baseline HbA1c value, treatment group, visit week, and treatment by visit week interaction. Unstructured covariance matrix was used; difference in least squares mean (LSM) = -0.11, 95% CI 2-sided [-0.31 to 0.10] — The estimation (LSM) is of the placebo-corrected change from baseline

2. Secondary Outcome: Change From Baseline in Fasting Serum Glucose at Week 24
Description: The average (mean) change from baseline in fasting serum glucose at Week 24 was analyzed.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Metformin | Ranolazine+Metformin
Number analyzed (Participants) | 171 | 176
mg/dL | -3 (44.7) | 3 (42.5)

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Serum Glucose at Week 24
Description: The average (mean) change from baseline in 2-hour postprandial serum glucose at Week 24 was analyzed.
  Mixed Meal Tolerance Test (MMTT) Full Analysis Set: randomized participants who received at least one dose of study treatment with a baseline and at least one postbaseline measurement of serum glucose at T=120 minutes during the MMTT, administered under fasting conditions, excluding participants with major eligibility protocol violations; analyzed based on the randomized treatment regardless of actual treatment received.
Time Frame: Baseline; Week 24
Population: Participants in the MMTT Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo+Metformin | Ranolazine+Metformin
Number analyzed (Participants) | 166 | 173
mg/dL | -4 (54.0) | 7 (58.2)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Arm/Group | Placebo+Metformin | Ranolazine+Metformin
Serious Adverse Events (participants affected / at risk) | 2/222 | 3/220
Other Adverse Events (participants affected / at risk) | 14/222 | 18/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Metformin (N=222) | Ranolazine+Metformin (N=220)
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Metformin (N=222) | Ranolazine+Metformin (N=220)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years